CLINICAL TRIAL: NCT01451892
Title: The Effect of Dance Therapy on the Functional Capacity of Patients With Advanced Obesity
Brief Title: Dance Therapy and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Principal Investigator, Lara Allet, Principal Investigator, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-072; 13DPD6_132361/1 (Other Grant/Funding Number: 13DPD6_132361/1)
Record Dates: First submitted 2011-10-05; First posted 2011-10-14 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: Obesity; dance; gait; balance; posture; dance therapy
MeSH Terms: conditions — Obesity | interventions — Dance Therapy; Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dance therapy (Experimental): overweight individuals participating in a patient education program for obese people combined with specific dance-therapy
  Interventions: Other: Dance Therapy
- Education (Active Comparator): overweight individuals participating in a patient education ambulatory program for obese people
  Interventions: Other: patient education

INTERVENTIONS:
Other: Dance Therapy — overweight individuals participating in a patient education program for obese people combined with specific dance-therapy
  Arms: Dance therapy
Other: patient education — overweight individuals participating in a patient education program
  Arms: Education

SUMMARY:
Title:

The effect of dance-therapy on the functional capacity, body image and quality of life of patients with advanced obesity

Project duration:

33 months (August 2010 to June 2013)

Clinical context:

Obesity has reached epidemic proportions. The gait and balance problems in obese people and the associated decreased functional capacity and risk of falling highlight the need to evaluate the benefits of specific treatments on these problems. Attention should be paid not only to metabolic management but also to the physical rehabilitation required in cases of advanced obesity.

Objectives:

The aim of this study is to evaluate the efficacy of dance-therapy on functional capacity (walking ability, postural control and physical activity level), body image and quality of life of patients with advanced obesity.

ELIGIBILITY:
Inclusion Criteria:

* Person with obesity (BMI ≥ 30)
* Aged > 18 years old
* Being able to walk 10 meters without a walking aid

Exclusion Criteria:

* Foot ulcer at the moment of data acquisition
* Orthopaedic, surgical or neurological (other than diabetic neuropathy ) problems which af-fect patient's gait
* Non diabetic neuropathy (Charcot, chronic alcohol consumption, thyroid dysfunction)
* Mental diseases interfering with group therapies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in comfortable gait speed | 0, 36 weeks, 6 months

SECONDARY OUTCOMES:
Change in functional capacities | 0, 36 weeks, 6 months
  * Change in cadence during normal gait(steps per minute)
  * Change in stride length during normal gait (meters)
  * Change in stride to stride variability during normal gait
  * Change in postural control: Displacement of the centre of pressure (COP) while standing on a stable and unstable surface
  * Change in functional parameters: Increase in maximal walking distance covered in 6 minutes (meters)
  * Change in required time to realize the Timed Up and Go Test (seconds)
  * Change in the Physical Activity Level and Total Energy expenditure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Allet L, Muller-Pinget S, Punt I, Edelsten C, Ballif A, Golay A, Pataky Z. Dance therapy combined with patient education improves quality of life of persons with obesity: A pilot feasibility study for a randomised controlled trial. Obes Res Clin Pract. 2017 Jan-Feb;11(1):79-87. doi: 10.1016/j.orcp.2016.03.005. Epub 2016 Apr 3. PMID 27053574